CLINICAL TRIAL: NCT02449096
Title: Operative Treatment of Complex Ankle Fractures: Comparison of the Results With and Without Ankle Arthroscopy-a Randomized Controlled Trial
Brief Title: Comparison of the Results of Complex Ankle Fractures Treated With and Without Ankle Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Mareen Braunstein, M.D., Dr. med. Mareen Braunstein, M.D., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117-15
Record Dates: First submitted 2015-04-07; First posted 2015-05-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures | interventions — Arthroscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ORIF group (Other): No arthroscope ORIF = Open reduction and internal fixation
  All Patients will be operated following a standardized protocol of our foot and ankle department:
  Posterior malleolus: ORIF of the posterior malleolus fractures will be performed using a one-third tubular plate in an antiglide-technique.
  Lateral malleolus: If the patients suffer a fracture of the posterior and lateral malleolus, a posterolateral approach will be performed. After posterior fracture fixation a lag screw and a one-third tubular plate will be used laterally. In special cases a locking plate will be used. If the patient only suffers a lateral malleolus fracture, we utilize the standard lateral incision.
  Medial malleolus: We perform a curved incision and two cannulated leg screws/tension wiring or locking plate for fixation.
  Syndesmotic complex: After all, the stability of the syndesmotic complex is tested and reduction will be performed if necessary.
  Interventions: Other: No arthroscope
- AORIF group (Active Comparator): Arthroscope AORIF = Arthroscopically assisted open reduction and internal fixation Our standard operative protocol is described above. Intervention: In case of randomization to the AORIF group, the arthroscopic procedure will be performed as the first step during the surgery before internal fixation. No distraction device will be used for the ankle. To avoid lesions of the cartilage and soft tissue, the joint will first be inflated with saline, and the portals will be created by blunt dissection. A 2.7mm, 30° arthroscope will be inserted into the ankle through a standard anteromedial portal. Fluid will be aspirated and the cavity filled with water. Afterwards the standard anterolateral portal will be performed in the same way. A standardized systematic examination as described by Ferkel and Fasulo will be performed to inspect the internal structures. At this stage loose bodies and disrupted ligaments extending into the joint will be removed.
  Interventions: Device: Arthroscope

INTERVENTIONS:
Device: Arthroscope — AORIF - arthroscopically assisted open reduction and internal fixation of acute ankle fractures
  Arms: AORIF group
Other: No arthroscope — ORIF - open reduction and internal fixation of acute ankle fractures
  Arms: ORIF group

SUMMARY:
Background: An anatomical reconstruction of ankle congruity is an important prerequisite in the operative treatment of acute ankle fractures. But, despite an anatomic reduction, patients suffer from residual problems like chronic pain, stiffness, persistent swelling and instability after these fractures. There is growing evidence, that this poor outcome is related to the concomitant traumatic intraarticular pathology. Therefore, supplementary ankle arthroscopy has been proposed in acute ankle fractures as it is a valuable tool to confirm the anatomic reposition and to further identify and manage associated intraarticular injuries. The arthroscopic treatment of these pathologies might result in a better outcome after complex ankle fractures. Nevertheless, until now, the vast majority of ankle fractures are managed by open procedures only. Still, indications for arthroscopically assisted open reduction and internal fixation (AORIF) are not clearly stated, and the effectiveness of AORIF compared with open reduction and internal fixation (ORIF) has not yet been determined for complex ankle fractures. In this context, only a prospective randomized study can sufficiently answer these open questions. Therefore, the investigators plan a randomized controlled trial intended to report the short-, midterm- and long-term follow-up of patients who underwent operative treatment of acute ankle fractures - with and without ankle arthroscopy.

Methods/Study design: The investigators will perform a randomized controlled trial evaluating the effect of AORIF compared to ORIF with a sample size of 40 patients per group. The investigators include patients with an acute ankle fracture after written informed consent. Primary outcome of the investigators' study is the difference of the AOFAS score (American Orthopedic Foot and Ankle Society) between the intervention (AORIF) and comparison (ORIF) group after a follow-up of 2 years. Several secondary outcome parameters will be assessed as well. Statistical analysis will be performed using a two-sided Student's t-test.

Discussion: Until today, there are only two randomized controlled trials evaluating the effect of open reduction and internal fixation (ORIF) compared to arthroscopically assisted open reduction and internal fixation (AORIF). Both studies only included patients with isolated fractures of the distal fibula at the level of the syndesmosis. These are the most simple fractures that are regularly treated operatively. Both studies documented a high incidence of intraarticular disorders in the AORIF group, but only one could show significant better results in the AORIF group. Moreover, several other studies could consistently demonstrate that the intraarticular damage is even more pronounced the more complex the fracture is. Consequently, a more distinctive effect of arthroscopy in complex fractures involving two malleoli or more has to be assumed when compared to these simple fractures.

DETAILED DESCRIPTION:
Acute ankle fractures are one of the leading pathologies disturbing ankle congruence. These fractures are extremely common with an incidence of 0.1-0.2% per year. The treatment of acute ankle fractures is determined by the classification of the injury based on radiographic findings. Operative treatment performing open reduction and internal fixation (ORIF) is the standard of care for unstable or dislocated ankle fractures. Anatomical realignment of the joint and restoration of ankle stability are the main goals of the operative treatment. Over the last decades the improved functional outcome has emphasized the importance of anatomic reconstruction. Nevertheless, successful anatomical reduction does not automatically lead to favorable clinical outcome. According to several studies, the mid- and long-term outcome following operative treatment of acute ankle fractures is often poor even though anatomical reconstruction of the joint has been achieved. Residual problems after acute ankle fractures include chronic pain, stiffness, recurrent swelling and instability. These problems occur despite the operative restoration of ankle congruence. There is growing evidence that the poor outcome might be mostly related to occult articular injuries involving cartilage and soft tissue damage. These intraarticular disorders have been shown to negatively affect the clinical results, but it is difficult to diagnose these intraarticular pathologies by physical examination, standard radiography or even CT-scans. In this context, many authors have well documented the value of ankle arthroscopy. Ankle arthroscopy is a standard minimally invasive technique that allows direct visualization of intraarticular structures without arthrotomy or malleolar osteotomy. In the last decades, it has become a safe and effective diagnostic and therapeutic procedure. In acute ankle fractures, arthroscopically assisted open reduction and internal fixation (AORIF) allows careful examination of the chondral aspects as well as the capsular and intraarticular ligaments. If necessary, the traumatic intraarticular pathologies can directly be addressed by removing loose bodies and ruptured ligaments extending into the joint, performing chondroplasty or micro fracturing if necessary. Furthermore, it allows a confirmation of the anatomic reduction without having any evidence that a supplementary ankle arthroscopy in acute ankle fracture treatment leads to a higher complication rate.

Until today, there are only two randomized controlled trials evaluating the effect of additional ankle arthroscopy. Both studies available comparing ORIF to AORIF included only patients with isolated fractures of the distal fibula at the level of the syndesmosis only. These are the most simple fractures that are regularly treated operatively. Thodarson et al. compared ORIF treatment of distal fibula fractures supplemented with or without ankle arthroscopy and found that 8 of 9 patients had articular damage to the talar dome in the arthroscopy group. Only minimal arthroscopic treatment was required and no outcome differences were noted after a mean follow-up of 21 months. Takao et al. documented an osteochondral lesion (OCL) in 74% in the arthroscopic group. In their study, the mean AOFAS score was significantly better when patients were treated arthroscopically. Moreover, several studies could consistently document, that the intraarticular damage is more pronounced the more complex the fracture is. Consequently, one must assume a more distinctive effect of arthroscopy in more complex fractures involving two malleoli or more - when compared to simple fractures.

Nevertheless, until now, the vast majority of ankle fractures are managed by open procedures only. Still, indications for AORIF are not clearly stated, and the effectiveness of AORIF compared with ORIF has not yet been determined for complex ankle fractures where the investigators would expect even better results as intraarticular lesions are more common in these fracture types. Moreover, the prognostic importance of traumatic articular lesions still remains unclear, although several studies suggest such injuries may be the source of functional deficits. Nevertheless, this concept seems to be intuitively comprehensible. In this context, only a prospective randomized study can sufficiently answer these open questions. Therefore, the investigators plan a randomized controlled trial intended to report the short-, midterm- and long-term follow-up of patients who underwent operative treatment of acute ankle fractures (AO A2, A3, B2, B3, C1-C3) - with and without ankle arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -65 years
* Acute ankle fracture (0-14 days) classified as AO type 44 A2, A3, B2, B3, C1-C3
* Written informed consent (patient is able to read and understand German language properly)

Exclusion Criteria:

* Patients under 18 years or over 65 years
* Patients who have acute infections, mental illnesses, high anesthesiological risk (ASA >3)
* Patients with expected incompliance
* Pregnant women, prisoners or patients under guardianship
* Acute ankle fracture classified as AO type 44 A1 or B1 fracture, pilon or plafond-variant injury
* Open fractures
* Fractures with radiologically detectable intraarticular lesions
* Patients without written informed consent

Men and women aged 18-65 years with an acute ankle fracture (AO 44 A2, A3, B2, B3, C1, C2, C3) according to the judgment of the surgeons of the foot and ankle team of our level I trauma center are enrolled in the trial. Each fracture will be evaluated and graded according to classification reported by AO Foundation (figure 1). Patients will be informed about our current investigation by detailed patient information. Only patients, who confirm the operative procedure, will be enrolled. To avoid misclassification, all radiographs will be evaluated by at least two of the three orthopedic surgeons. Disagreements will be resolved by consent. Only patients with a maximum interval of two weeks between injury and intervention must be included. All patients included must be able to understand the meaning of the trial and its consequences. Written informed consent is mandatory for trial inclusion. No additional investigation (clinical or radiographic investigation) will take place if the patient is included compared to patients who refuse inclusion. A list of inclusion and exclusion criteria can be found below. Patients will be excluded in case of open fractures or radiographically identified intraarticular lesions. Also, patients with a high risk of anesthesiology problems (i.e., ASA risk score > 3), acute infection, mental illness or low expected compliance will be excluded from trial participation. If patients issue a certain treatment preference, they will be excluded as well. Patients, who meet our inclusion criteria or any exclusion criteria, will be informed in detail. After written informed consent, patients will be randomized to one of the two study arms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
AOFAS (American Orthopedic Foot and Ankle Society) Score | 24 months (1-10 year follow-up anticipated)

SECONDARY OUTCOMES:
JSSF Score (Japanese Society of Surgery of the Foot) | 24 months (1-10 year follow-up anticipated)
Olerud and Molander Score | 24 months
Karlsson Score | 24 months
Tegner Activity Scale | 24 months
SF-12 Questionnaire | 24 months
Radiographic analysis | 24 months
Arthroscopic findings of intraarticular lesions | 24 months
Time to return to work/sports | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hans Polzer, M.D., Study Director — Munich University Clinic, Ludwig-Maximilians-University, Department of Trauma Surgery, Foot and Ankle Surgery, LMU, Munich
Locations (1):
- Ludwig Maximilians University, LMU, Munich, Munich, Bavaria, Germany

REFERENCES:
- [Background] Sorrento DL, Mlodzienski A. Incidence of lateral talar dome lesions in SER IV ankle fractures. J Foot Ankle Surg. 2000 Nov-Dec;39(6):354-8. doi: 10.1016/s1067-2516(00)80070-8. PMID 11131471
- [Background] Bonasia DE, Rossi R, Saltzman CL, Amendola A. The role of arthroscopy in the management of fractures about the ankle. J Am Acad Orthop Surg. 2011 Apr;19(4):226-35. doi: 10.5435/00124635-201104000-00007. PMID 21464216
- [Background] Hintermann B, Regazzoni P, Lampert C, Stutz G, Gachter A. Arthroscopic findings in acute fractures of the ankle. J Bone Joint Surg Br. 2000 Apr;82(3):345-51. doi: 10.1302/0301-620x.82b3.10064. PMID 10813167
- [Background] Aktas S, Kocaoglu B, Gereli A, Nalbantodlu U, Guven O. Incidence of chondral lesions of talar dome in ankle fracture types. Foot Ankle Int. 2008 Mar;29(3):287-92. doi: 10.3113/FAI.2008.0287. PMID 18348824
- [Background] Loren GJ, Ferkel RD. Arthroscopic assessment of occult intra-articular injury in acute ankle fractures. Arthroscopy. 2002 Apr;18(4):412-21. doi: 10.1053/jars.2002.32317. PMID 11951201
- [Background] Takao M, Ochi M, Uchio Y, Naito K, Kono T, Oae K. Osteochondral lesions of the talar dome associated with trauma. Arthroscopy. 2003 Dec;19(10):1061-7. doi: 10.1016/j.arthro.2003.10.019. PMID 14673447
- [Background] Takao M, Ochi M, Naito K, Uchio Y, Kono T, Oae K. Arthroscopic drilling for chondral, subchondral, and combined chondral-subchondral lesions of the talar dome. Arthroscopy. 2003 May-Jun;19(5):524-30. doi: 10.1053/jars.2003.50111. PMID 12724683
- [Background] Ono A, Nishikawa S, Nagao A, Irie T, Sasaki M, Kouno T. Arthroscopically assisted treatment of ankle fractures: arthroscopic findings and surgical outcomes. Arthroscopy. 2004 Jul;20(6):627-31. doi: 10.1016/j.arthro.2004.04.070. PMID 15241315
- [Background] Glazebrook MA, Ganapathy V, Bridge MA, Stone JW, Allard JP. Evidence-based indications for ankle arthroscopy. Arthroscopy. 2009 Dec;25(12):1478-90. doi: 10.1016/j.arthro.2009.05.001. PMID 19962076
- [Background] Thordarson DB, Bains R, Shepherd LE. The role of ankle arthroscopy on the surgical management of ankle fractures. Foot Ankle Int. 2001 Feb;22(2):123-5. doi: 10.1177/107110070102200207. PMID 11249221
- [Background] Takao M, Uchio Y, Naito K, Fukazawa I, Kakimaru T, Ochi M. Diagnosis and treatment of combined intra-articular disorders in acute distal fibular fractures. J Trauma. 2004 Dec;57(6):1303-7. doi: 10.1097/01.ta.0000114062.42369.88. PMID 15625464
- [Background] Leontaritis N, Hinojosa L, Panchbhavi VK. Arthroscopically detected intra-articular lesions associated with acute ankle fractures. J Bone Joint Surg Am. 2009 Feb;91(2):333-9. doi: 10.2106/JBJS.H.00584. PMID 19181977
- [Derived] Braunstein M, Baumbach SF, Regauer M, Bocker W, Polzer H. The value of arthroscopy in the treatment of complex ankle fractures - a protocol of a randomised controlled trial. BMC Musculoskelet Disord. 2016 May 12;17:210. doi: 10.1186/s12891-016-1063-2. PMID 27175917